CLINICAL TRIAL: NCT00592293
Title: Proton Radiation for the Treatment of Pediatric Bone and Non-Rhabdomyosarcoma Soft Tissue Sarcomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston Children's Hospital (Other); Dana-Farber Cancer Institute (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Torunn Yock, MD, Director, Pediatric Radiation Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-326; Other (Other Grant/Funding Number: program income on C06 CA059267)
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Non-rhabdomyosarcoma Soft Tissue Sarcoma; Bone Sarcoma
Keywords: proton beam radiation
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Beam Radiation (Experimental): Proton Beam Radiation
  Interventions: Radiation: Proton Beam Radiation

INTERVENTIONS:
Radiation: Proton Beam Radiation — Once per day, 5 days a week for a total of 4 to 6 weeks.

SUMMARY:
The main purpose of this study is to assess the short term and the long term side effects of proton beam radiation for pediatric bone and non-rhabdomyosarcoma soft tissue sarcomas.

DETAILED DESCRIPTION:
* Participants will receive radiation treatments once per day, 5 days a week for a total of 4 to 6 weeks, depending on how much total dose the tumor requires. The radiation doctor will see the participant once each week to monitor and record any side effects they may have from radiation treatment.
* A special device will be made for each participant to help them hold still during the treatment. This may either be a mask or foam cradle, depending on the area to be treated.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Non-Rhabdomyosarcoma Soft Tissue Sarcoma (NRSTS) or bone sarcoma
* Less than or equal to 30 years of age
* Patients must have been treated with a standardly accepted chemotherapy regimen if chemotherapy is indicated
* Patients must be willing to receive follow-up care for a minimum of five years after treatment at MGH and annual visits unless it is too difficult to return to MGH for follow-up care. In that event, the patient or guardian must be willing to have their outside medical information released in order to track the results of treatment
* They or their legal guardian must give their informed consent
* Timing of radiation may be according to concurrent protocol

Exclusion Criteria:

* Co-morbidities that would make the use of radiation too toxic to deliver safely, such as serious local injury of collagen vascular disease
* Patients who are pregnant
* Previous treatment with radiation therapy
* Concurrent adriamycin or gemcitabine chemotherapy is planned, unless on a concurrent protocol

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2006-10-24 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torunn Yock, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Beam Radiation
Started | 70
Completed | 69
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 70
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 12.8 [1.1 to 22.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 60
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence (Estimated Percentage of Participants) Who Developed Toxicities Following Radiation Treatment
Description: Cumulative incidence (percent of participants and 95% confidence intervals) who experienced a grade 3, 4, or 5 late toxicity. Late complications are defined as the delayed effects attributable to radiation which occur > 90 days following completion of radiation.
Time Frame: 5 years from the completion of radiation treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 70
percentage of participants | 17.7 [9.7 to 28.8]
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; Cumulative incidence = 17, 95% CI 2-sided [9.1 to 27.6]

2. Primary Outcome: Local Control
Description: Rates of local control using proton radiotherapy. Local control is the lack of tumor recurrence in and or near the area where the primary tumor occurred.
Time Frame: 5 years from the start of radiation treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 70
percentage of participants | 87.1 [78.1 to 93.7]
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; Percent Survival, Local Control = 87.1, 95% CI 2-sided [78.1 to 93.7]

3. Secondary Outcome: Dosimetric Comparison
Description: Comparison of Dose distribution to tumor and surrounding normal structures using Dose-Volume Histograms (DVH) generated from the proton plan used to treat the patient and the photon plan generated for comparison purposes.
Time Frame: 5 years
Population: Data were not collected and this outcome was not analyzed. DVH's were not generated for these patients. Data will not be collected in the future. The decision not to generate photon/proton contours DVH's was at the discretion of the dosimetrist/treating physician.
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years following the completion of treatment, mean of 9.1 years
Description: Acute toxicity will be scored at weekly status check visits by the radiation oncology nurse or doctor. In addition, acute toxicity will be scored at least one time within the 3 months following completion of radiation therapy. Version 3.0. Late toxicity is to be scored on a yearly follow-up basis for at least five years. Toxicities and will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0.
Arm/Group | Proton Beam Radiation
All-Cause Mortality (participants affected / at risk) | 17/69
Serious Adverse Events (participants affected / at risk) | 8/69
Other Adverse Events (participants affected / at risk) | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Beam Radiation (N=69)
Myelodysplastic Syndrome (MDS) (Blood and lymphatic system disorders) | 1
Venoocclusive disease (Hepatobiliary disorders) | 1
Staphylocaccus bacteremia (Infections and infestations) | 1
Leukemia (AML) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelet count decreased (Investigations) | 1
Subglottic stenosis, tracheotomy (Respiratory, thoracic and mediastinal disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Beam Radiation (N=69)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 3
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 4
Hearing-other (Ear and labyrinth disorders) | 4
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 26
Leukocytes (Blood and lymphatic system disorders) | 30
Lymphopenia (Blood and lymphatic system disorders) | 30
Neutrophils (Blood and lymphatic system disorders) | 29
Platelets (Blood and lymphatic system disorders) | 27
Fatigue (General disorders) | 55
Fever w/o neutropenia (General disorders) | 1
Sweating (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 13
Bruising (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 22
Hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 65
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Skin-other (Skin and subcutaneous tissue disorders) | 6
Telangiectasia (Skin and subcutaneous tissue disorders) | 6
Wound - non-infectious (Skin and subcutaneous tissue disorders) | 1
ACTH deficiency (Endocrine disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 3
Endocrine-other (Endocrine disorders) | 2
Gonadotropin secretion abnormality (Endocrine disorders) | 4
Growth hormone secretion abnormality (Endocrine disorders) | 5
Hot flashes (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 8
Anorexia (Gastrointestinal disorders) | 25
Constipation (Gastrointestinal disorders) | 3
Dehydration (Gastrointestinal disorders) | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 6
Esophagitis (Gastrointestinal disorders) | 7
GI-other (Gastrointestinal disorders) | 4
Muco/stomatitis (symptom) pharynx (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 11
Muco/stomatitis by exam, pharynx (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Obstruction, small bowel NOS (Gastrointestinal disorders) | 1
Salivary (Gastrointestinal disorders) | 1
Stenosis (incl anastomotic) pharynx (Gastrointestinal disorders) | 1
Taste disturbance (Gastrointestinal disorders) | 2
Teeth (Gastrointestinal disorders) | 2
Teeth development (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Growth velocity reduction (General disorders) | 2
Short stature (General disorders) | 2
Spine kyphosis/lordosis (Musculoskeletal and connective tissue disorders) | 4
Hemorrhage-other (General disorders) | 3
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 6
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pharynx, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Infection w/ unk ANC sinus (Infections and infestations) | 1
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 1
Infection-other (Infections and infestations) | 6
AST, SGOT (Metabolism and nutrition disorders) | 2
Bilirubin (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Bone: spine-scoliosis (Musculoskeletal and connective tissue disorders) | 5
Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 4
Extremity upper (function) (Musculoskeletal and connective tissue disorders) | 1
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1
Fibrosis-cosmesis (Musculoskeletal and connective tissue disorders) | 2
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Joint-function (Musculoskeletal and connective tissue disorders) | 4
Lumbar spine-range of motion (Musculoskeletal and connective tissue disorders) | 1
Muscular/skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 10
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 17
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic left-side muscle weak (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic upper extr muscle weak (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Agitation (Psychiatric disorders) | 1
Cognitive disturbance (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 3
Memory impairment (Psychiatric disorders) | 1
Neurologic-other (Psychiatric disorders) | 3
Neuropathy-motor (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 7
Speech impairment (Psychiatric disorders) | 1
Cataract (Eye disorders) | 2
Dry eye syndrome (Eye disorders) | 4
Eyelid dysfunction (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Ocular-other (Eye disorders) | 7
Optic disc edema (Eye disorders) | 1
Tearing (Eye disorders) | 5
Vision-blurred (Eye disorders) | 1
Vision-photophobia (Eye disorders) | 1
Skin, pain (General disorders) | 1
Throat/pharynx/larynx, pain (General disorders) | 6
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 2
FEV1 (Respiratory, thoracic and mediastinal disorders) | 1
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 6
Obstruction, airway-pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 8
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 5
Bladder spasms (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 1
Obstruction-ureteral (Renal and urinary disorders) | 1
Renal/GU-other (Renal and urinary disorders) | 4
Urinary frequency/urgency (Renal and urinary disorders) | 5
Irregular menses (Reproductive system and breast disorders) | 4
Libido (Reproductive system and breast disorders) | 1
Sexual/Reproductive function-Other (Reproductive system and breast disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Vascular-Other (Specify) (Vascular disorders) | 1
Edema head and neck (General disorders) | 4
Edema limb (General disorders) | 2
Lymphatics-other (General disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 5
Back, pain (Musculoskeletal and connective tissue disorders) | 12
Buttock, pain (Musculoskeletal and connective tissue disorders) | 3
Dental/teeth/peridontal, pain (Gastrointestinal disorders) | 3
External ear, pain (Ear and labyrinth disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 4
Eye, pain (Eye disorders) | 2
Face, pain (General disorders) | 2
Head/headache (Nervous system disorders) | 7
Middle ear, pain (Ear and labyrinth disorders) | 2
Neck, pain (Musculoskeletal and connective tissue disorders) | 2
Oral cavity, pain (Gastrointestinal disorders) | 1
Oral gums, pain (Gastrointestinal disorders) | 1
Pain-other (General disorders) | 8
Pelvic, pain (Reproductive system and breast disorders) | 5
Scalp, pain (Skin and subcutaneous tissue disorders) | 1
Skin, pain (Skin and subcutaneous tissue disorders) | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes